CLINICAL TRIAL: NCT06063668
Title: Serum Autotaxin as a Potential Biomarker in Systemic Lupus Erythematosus Patients and Its Relation to Disease Activity.
Brief Title: Autotaxin as Abiomarker in Systemic Lupus Erythematosus Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Mohamed Abd-Elrazik Ahmed, Resident doctor, Assiut University
Other Study IDs: Autotaxin in sle
Record Dates: First submitted 2023-09-24; First posted 2023-10-02 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: SLE (Systemic Lupus)
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients: SLE patients
- controls: healthy controls

SUMMARY:
* Estimation of the serum ATX level in SLE patients in comparison to healthy subjects.
* Evaluation of the relation of serum ATX level with disease activity and different clinical manifestation in SLE patients

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic multisystem autoimmune inflammatory disease with unknown etiology . However, several genetic, immunological and environmental factors play a role in the etiopathogenesis of SLE . During the disease course, patients may be presented with diverse clinical manifestations (mucocutaneous, articular, neurological, or renal manifestations) . Anti-nuclear antibodies(ANA), anti- double stranded DNA (ds-DNA)and anti smith(SM) antibodies are common biomarkers of SLE. However the sensitivity and specificity of the current biomarkers are not ideal that the diagnosis of SLE can be missed .

Lysophospholipids are phospholipids with only one fatty acid chain, such as lysophosphatidic acid (LPA) and lysophosphatidylserine. Autotaxin (ATX), one of the enzymes that catalyze the formation of Lysophospholipid, is mainly responsible for the production of LPA in blood . Tumor necrosis factor (TNF), interleukin-6 (IL-6), and type I interferons, have been reported to induce the expression of ATX . ATX was reported recently as potential biomarkers of various diseases (serum ATX in malignancy and chronic hepatitis C, while in acute myocardial infarction ATX was overexpressed in cardiac tissue and in the synovium of rheumatoid arthritis patients) . Several studies have reported that serum ATX concentrations were higher in females than in males . The mRNA expression of ATX was found to be significantly induced by estrogen . There is growing evidence that ATX may play a role in the pathogenesis of SLE. Few recent studies have reported that serum ATX level can be a possible novel biomarker and key molecule in SLE .

ELIGIBILITY:
Inclusion Criteria:

* Patients who will be diagnosed as SLE according to the 2012 systemic lupus international collaborating clinics (SLICC) criteria .
* SLE Patients older than 18 years old.

Exclusion Criteria:

* SLE Patients younger than 18 years old.
* Patients with other rheumatic diseases or overlap syndromes.
* Patients with malignancy.
* Patients with chronic hepatitis C.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: SLE patients fullfilling the 2012 systemic lupus international collaborating clinics (SLICC) criteria ,older than 18 years old with no other rheumatic diseases or malignancy.
  Controls are healthy controls .
Sampling Method: Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Serum ATX level in SLE patients in comparison to healthy controls. | 2 years
  Measure ATX level in serum of sle patients and compare it with ATX level in serum of healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Nada Mohamed Gamal Abd-Elaleem, Ass. Prof, Study Chair — Assiut University; Maha Sayed Ibrahim Abdelrahman, Lecturer, Study Chair — Assiut University

REFERENCES:
- [Result] Tsuchida Y, Shoda H, Sawada T, Fujio K. Role of autotaxin in systemic lupus erythematosus. Front Med (Lausanne). 2023 Apr 4;10:1166343. doi: 10.3389/fmed.2023.1166343. eCollection 2023. PMID 37122329
- [Result] Tsuchida Y, Shoda H, Nakano M, Ota M, Okamura T, Yamamoto K, Kurano M, Yatomi Y, Fujio K, Sawada T. Autotaxin is a potential link between genetic risk factors and immunological disturbances of plasmacytoid dendritic cells in systematic lupus erythematosus. Lupus. 2022 Nov;31(13):1578-1585. doi: 10.1177/09612033221128494. Epub 2022 Sep 22. PMID 36134766
- [Result] Cojocaru M, Cojocaru IM, Silosi I, Vrabie CD. Manifestations of systemic lupus erythematosus. Maedica (Bucur). 2011 Oct;6(4):330-6. PMID 22879850
- [Result] Magkrioti C, Galaris A, Kanellopoulou P, Stylianaki EA, Kaffe E, Aidinis V. Autotaxin and chronic inflammatory diseases. J Autoimmun. 2019 Nov;104:102327. doi: 10.1016/j.jaut.2019.102327. Epub 2019 Aug 28. PMID 31471142
- [Result] Iwata Y, Kitajima S, Yamahana J, Shimomura S, Yoneda-Nakagawa S, Sakai N, Furuichi K, Ogura H, Sato K, Toyama T, Yamamura Y, Miyagawa T, Hara A, Shimizu M, Ohkawa R, Kurano M, Yatomi Y, Wada T. Higher serum levels of autotaxin and phosphatidylserine-specific phospholipase A1 in patients with lupus nephritis. Int J Rheum Dis. 2021 Feb;24(2):231-239. doi: 10.1111/1756-185X.14031. Epub 2020 Dec 11. PMID 33314787
- [Result] Gladman DD, Ibanez D, Urowitz MB. Systemic lupus erythematosus disease activity index 2000. J Rheumatol. 2002 Feb;29(2):288-91. PMID 11838846
- [Result] Tan EM. Antinuclear antibodies: diagnostic markers for autoimmune diseases and probes for cell biology. Adv Immunol. 1989;44:93-151. doi: 10.1016/s0065-2776(08)60641-0. No abstract available. PMID 2646863
- [Result] Yu H, Nagafuchi Y, Fujio K. Clinical and Immunological Biomarkers for Systemic Lupus Erythematosus. Biomolecules. 2021 Jun 22;11(7):928. doi: 10.3390/biom11070928. PMID 34206696
- [Result] Masuda A, Nakamura K, Izutsu K, Igarashi K, Ohkawa R, Jona M, Higashi K, Yokota H, Okudaira S, Kishimoto T, Watanabe T, Koike Y, Ikeda H, Kozai Y, Kurokawa M, Aoki J, Yatomi Y. Serum autotaxin measurement in haematological malignancies: a promising marker for follicular lymphoma. Br J Haematol. 2008 Oct;143(1):60-70. doi: 10.1111/j.1365-2141.2008.07325.x. Epub 2008 Aug 15. PMID 18710386
- [Result] Tokuhara Y, Kurano M, Shimamoto S, Igarashi K, Nojiri T, Kobayashi T, Masuda A, Ikeda H, Nagamatsu T, Fujii T, Aoki J, Yatomi Y. A New Enzyme Immunoassay for the Quantitative Determination of Classical Autotaxins (ATXalpha, ATXbeta, and ATXgamma) and Novel Autotaxins (ATXdelta and ATXepsilon). PLoS One. 2015 Jun 17;10(6):e0130074. doi: 10.1371/journal.pone.0130074. eCollection 2015. PMID 26083365
- [Result] Zhang G, Cheng Y, Zhang Q, Li X, Zhou J, Wang J, Wei L. ATX-LPA axis facilitates estrogen-induced endometrial cancer cell proliferation via MAPK/ERK signaling pathway. Mol Med Rep. 2018 Mar;17(3):4245-4252. doi: 10.3892/mmr.2018.8392. Epub 2018 Jan 8. PMID 29328374
- [Result] Petri M, Orbai AM, Alarcon GS, Gordon C, Merrill JT, Fortin PR, Bruce IN, Isenberg D, Wallace DJ, Nived O, Sturfelt G, Ramsey-Goldman R, Bae SC, Hanly JG, Sanchez-Guerrero J, Clarke A, Aranow C, Manzi S, Urowitz M, Gladman D, Kalunian K, Costner M, Werth VP, Zoma A, Bernatsky S, Ruiz-Irastorza G, Khamashta MA, Jacobsen S, Buyon JP, Maddison P, Dooley MA, van Vollenhoven RF, Ginzler E, Stoll T, Peschken C, Jorizzo JL, Callen JP, Lim SS, Fessler BJ, Inanc M, Kamen DL, Rahman A, Steinsson K, Franks AG Jr, Sigler L, Hameed S, Fang H, Pham N, Brey R, Weisman MH, McGwin G Jr, Magder LS. Derivation and validation of the Systemic Lupus International Collaborating Clinics classification criteria for systemic lupus erythematosus. Arthritis Rheum. 2012 Aug;64(8):2677-86. doi: 10.1002/art.34473. PMID 22553077
- [Result] Stoll T, Seifert B, Isenberg DA. SLICC/ACR Damage Index is valid, and renal and pulmonary organ scores are predictors of severe outcome in patients with systemic lupus erythematosus. Br J Rheumatol. 1996 Mar;35(3):248-54. doi: 10.1093/rheumatology/35.3.248. PMID 8620300